CLINICAL TRIAL: NCT06838338
Title: A Phase Ib, Open Lable, Clinical Trial of JAB-21822 Combined With Second Line Chemotherapy and Bevacizumab for Metastatic Colorectal Cancer With KRAS G12C Mutation
Brief Title: JAB-21822 Combined With Chemotherapy and Bevacizumab in Second-line KRAS G12C CRC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jian Li (Other)
Responsible Party: Sponsor-Investigator, Jian Li, Chief Physician, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JAB-21822-CRC003
Record Dates: First submitted 2024-09-25; First posted 2025-02-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JAB-21822 and second-line standard chemotherapy with bevacizumab (Experimental): Patients receive JAB-21822 combined with chemotherapy with bevacizumab as the second-line treatment until disease progression or intolerable toxicity
  Interventions: Drug: JAB-21822; Drug: standard second-line chemotherapy; Drug: Bevacizumab

INTERVENTIONS:
Drug: JAB-21822 — Tablet, oral, 800 mg/QD, until PD or intolerable toxicity
Drug: standard second-line chemotherapy — The second line standard chemotherapy regimen recommended by clinical practice
  Other Names: FOLFIRI, FOLFOX
Drug: Bevacizumab — 5mg/kg every two weeks (according to the assessment by investigator)

SUMMARY:
KRAS is a common genetic mutation in tumors, and CRC is one of the tumors with a high KRAS mutation rate. The anti-tumor activity of KRAS G12C inhibitors combined with anti-EGFR anti-bodies have been proven in patients with advanced colorectal cancer, and one of them was approved for patients who have previously received standard treatment. However, Chinese patients still do not have access to these drugs. This study is to determine the efficacy and safety of KRAS G12C inhibitor JAB-21822 in combination with the second-line standard chemotherapy and bevacizumab in advanced colorectal cancer failed to standard therapy in Chinese population.

DETAILED DESCRIPTION:
The study is aimed for patients with histologically confirmed advanced metastatic colorectal cancer with KRAS G12C mutation, patients enrolled will treated with JAB-21822 combined with standard second-line chemotherapy and bevacizumab until disease progression or intolerable toxicity or patient-initiated withdrawal from the study. Enrolled patients will undergo imaging assessments at baseline and every 6 weeks during the treatment period, the anti-tumor efficacy will be evaluated by the investigator according to RECIST v1.1. Safety assessment included vital signs, haematology, blood biochemistry and urinalysis and will be monitored regularly during the study period during treatment. Any discomfort experienced by the patients after administration of the drug will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Histologically (or cytologically) confirmed, unresectable metastatic colorectal cancer.
* KRAS G12C mutation.
* At least one measurable disease per RECIST v1.1; assessed within 28 days before first dose.
* Subject have withdrawn from the first-line chemotherapy due to disease progression or unacceptable toxicity; if first-line chemotherapy and maintenance therapy were received, disease progression must within three months; first-line chemotherapy regimens do not limit the use of antiangiogenic agents.
* Adequate bone marrow, liver and renal function.
* ECOG performance status 0-1.
* Informed consent has been signed.

Exclusion Criteria:

* Patients have received KRAS G12C inhibitors.
* Patients have received a first-line treatment, which include fluoropyrimidine, oxaliplatin and irinotecan.
* Patients who are pregnant or breastfeeding.
* Life expectancy of less than 3 months.
* Patients who had major surgery or significant trauma within 4 weeks prior to the first blood sample collection during the screening period, or expected to require major surgery during the study period.
* Patients with active ulcers and gastrointestinal bleeding.
* Prior history of interstitial lung disease or non-infectious pneumonia; history of active tuberculosis.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
* Patients with clinically diagnosed autoimmune disease; HIV, HCV positive; HBV-DNA beyond the normal range of the laboratory; Acute CMV infection.
* Patients with active central nervous system metastases requiring treatment.
* Patients with other malignancies within five years.
* Assessed by the investigator, patients who are unable or unwilling to comply with the requirements of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Time Frame: up to 1year
  The percentage of patients with total number of Complete Response (CR) + total number of Partial Response (PR) per RECIST v1.1

SECONDARY OUTCOMES:
Overall Survival (OS) | Time Frame: up to 1 year
  Defined as the time from date of study treatment to death due to any cause.
Progression-free Survival (PFS) | Time Frame: up to 1 year
  Defined as the time from date of study treatment to disease progression radiological/clinical or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | Time Frame: up to 1 year
  Defined as the percentage of patients whose best response are not Progressive Disease (PD) according to RECIST v1.1.
Duration of Response (DOR) | Time Frame: up to 1 year
  Defined as the time between the first assessment of the tumor as a CR or PR and the first assessment as disease progression (PD) or death from any cause.
Rate of treatment-related adverse events | Time Frame: up to 1 year
  Number of patients with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobio Pharmaceuticals, Study Director — Jacobio Pharmaceuticals
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University Cancer Hospital (Inner Mongolia Campus)/Afffliated Cancer Hospital of Inner Mongolia Medical University, Hohhot
  - Fudan University Shanghai Cancer Center, Shanghai